CLINICAL TRIAL: NCT06130501
Title: IMBUE RETAIN: Transcutaneous Auricular Neurostimulation (tAN) for Patients With Co-occurring Posttraumatic Stress Disorder (PTSD) and Opioid Use Disorder Starting Buprenorphine Therapy
Brief Title: tAN for PTSD and OUD in Buprenorphine Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Spark Biomedical, Inc. (Industry)
Responsible Party: Principal Investigator, Joel G Sprunger, PhD, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1UG3DA059409-01 (NIH)
Record Dates: First submitted 2023-10-26; First posted 2023-11-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Posttraumatic Stress Disorder; Opioid Use Disorder
Keywords: feasibility; medication for opioid use disorder (buprenorphine); treatment retention; transcutaneous auricular neurostimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The Research Coordinator, Project Manager, and Site PI will be unblinded so that the participant receives the appropriate device for their assigned treatment condition, they are able to provide technical support, and give the participant feedback on their dose compliance throughout the study. The participant, all outcomes assessors, and the participant's buprenorphine care provider will be blind to condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tAN (Experimental): Participants receive active tAN with the Sparrow Ascent device from Spark Biomedical (Dallas, TX).
  Interventions: Device: Sparrow Ascent tAN
- Active Sham (Sham Comparator): Participants receive the active sham version of the Sparrow Ascent device that limits stimulation to trigeminal innervation only and at a charge that is approximately 1000x lower than the active tAN condition.
  Interventions: Device: Sparrow Ascent Active Sham

INTERVENTIONS:
Device: Sparrow Ascent tAN — The Sparrow Ascent device from Spark Biomedical (Dallas, TX), applies stimulation frequencies of 15 Hz at the cymba concha (vagal innervation) and 100 Hz anterior to the tragus (trigeminal innervation). Both tAN and active sham conditions have square biphasic waveforms with identical pulse widths of 250 µs separated by a 125 µs interval between pulses. Stimulation is applied using a duty cycle of 5-minutes ON and 10 seconds OFF. The stimulation intensities (mA) will be programmed for each individual based on the highest amplitude for each channel that is both comfortable and perceptible. Patients using the device may alter the intensity of stimulation at these sites using the Patient Controller to achieve the desired effect.
  Other Names: Sparrow Ascent System; Sparrow Ascent tAN System
  Arms: Active tAN
Device: Sparrow Ascent Active Sham — The Sparrow Ascent Active Sham is a modified version of the Sparrow Ascent tAN System that has been designed to provide sub-therapeutic stimulation to the trigeminal nerve only and no stimulation to the vagus nerve. The trigeminal nerve will receive 1 Hz stimulation at the temporomandibular region at an amplitude that is comfortable and perceptual. The pulse duration will be set to a value that does not exceed 250 μs in a square biphasic waveform. The patient controller device for the active sham will give the appearance that stimulation is being applied at both vagal and trigeminal electrode sites.
  Arms: Active Sham

SUMMARY:
The goal of this research study supported by the HEAL Initiative (https://heal.nih.gov) is to investigate the effects transcutaneous auricular neurostimulation (tAN), as delivered through the Sparrow Ascent device, on helping people with co-occurring posttraumatic stress disorder (PTSD) and opioid use disorder (OUD) start and continue buprenorphine treatment. The main questions it aims to answer are:

* Does the tAN help participants with OUD and PTSD remain in buprenorphine therapy for three months after starting use of the device (i.e., randomization to treatment condition)?
* Do participants find the Sparrow Ascent device to be acceptable and use it?
* Do participants find the Sparrow Ascent device to be tolerable and comfortable to use?
* Do participants find the Sparrow Ascent device to be easy to use with their buprenorphine therapy?
* Do participants follow the minimum recommended dose schedule for the Sparrow Ascent device most of the time?

Participants will complete a baseline assessment to make sure that they are eligible to participate in the study. The assessment captures information about demographics, substance use and treatment history, opioid withdrawal symptoms and craving, difficult life experiences and PTSD symptoms, mental health and treatment history, quality of life, and recovery resources. After the assessment is complete and the participant has been inducted on buprenorphine as part of standard care, they are randomized to one of two treatment conditions: active tAN and placebo. Participants are trained on how to use the device and return for 12 weekly research visits to check on recent substance use and craving, PTSD symptoms, and their experience using the device. After 12 weeks of using the device, participants will complete a post-active treatment assessment that is nearly identical to the baseline assessment to see if there have been changes in these areas. Researchers will access the medical record to determine whether there is a current prescription for buprenorphine at three months and six months after randomization.

DETAILED DESCRIPTION:
Supported by the HEAL Initiative (https://heal.nih.gov), the overall UG3/UH3 phased project will test transcutaneous auricular neurostimulation (tAN) to the trigeminal and vagus nerves via the Sparrow Ascent device as an adjunct intervention to improve retention in buprenorphine treatment (BUP) for patients with co-occurring opioid use disorder and posttraumatic stress disorder. The specific objectives of the UG3 project are to:

1. conduct a pilot randomized, active sham-controlled test of transcutaneous auricular neurostimulation (tAN) with the Sparrow Ascent device to determine its acceptability, tolerability, feasibility, and adherence in patients with OUD and PTSD starting buprenorphine (BUP) therapy;
2. submit progress for review regarding study milestones and go/no-go criteria for approval of the UH3 phase; and
3. complete FDA pre-submission for FDA input on proposed UH3 protocols to expand Sparrow Ascent's indication for PTSD symptoms.

Approximately twenty adults diagnosed with opioid use disorder and posttraumatic stress disorder initiating buprenorphine treatment will complete a baseline assessment of substance use and mental health diagnostic measures before being randomized into the study. Participants randomized to the active tAN condition will receive therapeutic stimulation to the trigeminal and vagus nerves through the Sparrow Ascent earpiece when they activate their Patient Controller. Participants randomized to the active sham condition will receive only stimulation on the trigeminal nerve at a level that can be felt but is well below any therapeutic effect. All participants will receive identical training for the Sparrow Ascent device and the only difference will be the condition-dependent programming of their Patient Controllers. Participants begin using the Sparrow Ascent device within 28 calendar days of buprenorphine induction. For the next 12 weeks, as they continue through standard buprenorphine treatment, participants will independently administer stimulation at or above a recommended dosage schedule that decreases in frequency every four weeks during the active participation period (i.e., Weeks 1-4, 5-8, 9-12). Device usage logs will be downloaded and assessed at weekly research visits throughout the active participation period to determine device adherence and provide feedback and assistance, if needed. After 12 weeks of device usage, participants return their device and complete a post-assessment that repeats many of the baseline assessments to determine changes from baseline. Buprenorphine treatment retention (primary outcome) at three months and six months (secondary outcome) post-randomization will be extracted from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65.
* Patient seeking buprenorphine therapy (BUP) for opioid use disorder and able to be randomized within 28 calendar days of induction on BUP.
* Meets Diagnostic and Statistical Manual - 5 (DSM-5) diagnostic criteria for moderate to severe opioid use disorder with induction on buprenorphine. This includes volunteers who have taken buprenorphine in the past and are re-starting, are currently receiving non-buprenorphine medication for opioid use disorder, or have taken non-buprenorphine medication for opioid use disorder in the past and are transitioning to buprenorphine therapy for the first time.
* Meets DSM-5 diagnostic criteria for posttraumatic stress disorder (PTSD).
* Is able to understand the study, and having understood, provide written informed consent in English.
* Provides permission to extract data from the participant's electronic medical record.

Exclusion Criteria:

* Unable to provide sufficient contact information (must provide at least two reliable indicators).
* Volunteers who will not undergo induction on BUP within the eligibility window for randomization.
* Volunteers who intend to, or will receive, inpatient substance use disorder (SUD) care at the time of randomization. Volunteers receiving inpatient detoxification care at the time of screening or baseline assessment are eligible if they will no longer be receiving inpatient care when they would be randomized for the study.
* Volunteers actively participating in evidence-based psychotherapy for PTSD (e.g., Prolonged Exposure, Cognitive Processing Therapy, etc.).
* Volunteers who will not have been stable on medications that affect PTSD (i.e., sertraline, paroxetine, venlafaxine, prazosin, or trazodone) for at least four weeks before they could be randomized.
* Volunteer presents current evidence of an uncontrolled and/or clinically significant medical or psychiatric condition that will impact their ability to comply with the study requirements or would make their study participation unsafe. This includes unmedicated bipolar disorder with a manic episode in the past month or unmedicated psychotic disorder.
* Volunteer has a history of epileptic seizure.
* Volunteer has a history of neurological disorder or traumatic brain injury with significant lasting effects (e.g., memory problems, emotional changes, behavioral changes).
* Volunteer had a suicide attempt leading to hospital admission in the past month or suicidal ideation with a plan and intent to act upon it in the past month.
* Volunteer has the presence of devices (e.g., pacemakers, cochlear prosthesis, neurostimulators).
* Volunteer has abnormal ear anatomy or an ear infection is present.
* Volunteer is pregnant or lactating.
* Volunteers of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study's active participation period (i.e., 12 weeks following randomization).
* Volunteer has any other significant medical or psychosocial problems that, in the opinion of the investigator, would potentially cause harm to the participant, impact their ability to participate, or influence the results of the project's trial. These include circumstances such as impending incarceration, moving out of the area, or a general history of noncompliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
3-month Buprenorphine (BUP) Retention | 3 months post-randomization
  3-month BUP retention, operationalized as a current BUP prescription at the time of data extraction (retained/not retained), will be examined by observing the proportion of participants who are retained in BUP therapy at 3 months post-randomization.

SECONDARY OUTCOMES:
Device Acceptability | 3 months post-randomization
  The proportion of participants registering use of the device.
Device Tolerability | 3 months post-randomization
  The proportions of participants endorsing that the device caused pain or discomfort to the ear, discontinue the study due to a device-related Adverse Event (AE), and any device-related Serious Adverse Events (SAEs).
Device Feasibility - Patient Ease of Use | 3 months post-randomization
  The proportion of participants who endorse that the device was easy to use as measured by the Device Usability Questionnaire using a five-item ordinal scale ranging from Strongly disagree to Strongly agree.
Device Feasibility - Patient Helpfulness | 3 months post-randomization
  The proportion of participants who endorse that the device helped them take their buprenorphine as prescribed as measured by the Device Usability Questionnaire using a five-item ordinal scale ranging from Strongly disagree to Strongly agree.
Device Feasibility - Patient Value | 3 months post-randomization
  The proportion of participants who endorse that the device is valuable for people with PTSD and OUD taking buprenorphine as measured by the Device Usability Questionnaire using a five-item ordinal scale ranging from Strongly disagree to Strongly agree.
Device Feasibility - Provider Helpfulness | 3 months post-randomization
  The proportion of provider reports of patient device usage endorsing that the device helped their participants take their buprenorphine as prescribed as measured by the Provider Feedback Questionnaire using a five-item ordinal scale ranging from Strongly disagree to Strongly agree.
Device Feasibility - Provider Utility | 3 months post-randomization
  The proportion of provider reports of patient device usage endorsing that the device has utility as an adjunct to buprenorphine therapy as measured by the Provider Feedback Questionnaire using a five-item ordinal scale ranging from Strongly disagree to Strongly agree.
Device Feasibility - Provider Value | 3 months post-randomization
  The proportion of provider reports of patient device usage endorsing that the device has value as a treatment option for patients with PTSD and OUD taking buprenorphine as measured by the Provider Feedback Questionnaire using a five-item ordinal scale ranging from Strongly disagree to Strongly agree.
Device Feasibility - Provider Barrier | 3 months post-randomization
  The proportion of provider reports of patient device usage endorsing that the device does not make it harder for their participant to take their medication as measured by the Provider Feedback Questionnaire using a five-item ordinal scale ranging from Strongly disagree to Strongly agree.
Device Adherence | 3 months post-randomization
  The proportion of participants who meet or exceed the minimum dosing schedule for at least 75% (9 of 12) weekly research visits.
Buprenorphine Medication Compliance | 3 months post-randomization
  The proportions of weekly research visits with a positive result for buprenorphine in the urine drug test and self-reported buprenorphine administration as prescribed.
Substance Use | 3 months post-randomization
  The proportions of weekly research visits with self-reported non-prescribed substance use (e.g., opioid use, stimulant use) as measured by the Timeline Follow-back Method and positive urine drug test results.
PTSD Symptom Severity - Self Rated | 3 months post-randomization
  Mean change in PTSD Checklist for DSM-5 (PCL-5) symptom severity scores from baseline to post-treatment assessment. PCL-5 scores range from 0 - 80 with a higher score indicating more severe trauma-related distress due to PTSD symptoms.
PTSD Symptom Severity - Clinician Rated | 3 months post-randomization
  Mean change in Clinician-administered PTSD Scale for DSM-5 (CAPS-5) symptom severity scores from baseline to post-treatment assessment. CAPS-5 scores range from 0 - 80 with a higher score indicating more severe trauma-related distress due to PTSD symptoms.
PTSD Remission Status | 3 months post-randomization
  Change in PTSD diagnostic status according to the Clinician-administered PTSD Scale for DSM-5 (CAPS-5).
Opioid Withdrawal Symptom Severity - Self Rated | 3 months post-randomization
  Mean change in self-reported opioid withdrawal symptom severity on the 10-item Short Opiate Withdrawal Scale - Gossop (SOWS-Gossop). Participants rate each item on a scale ranging from 0 (None) to 3 (Severe). The total scale score ranges between 0 - 30, with higher scores indicating more severe withdrawal symptoms.
Opioid Withdrawal Symptom Severity - Observer Rated | 3 months post-randomization
  Mean change in observer-rated severity on the 11-item Clinical Opiate Withdrawal Scale (COWS). The total score on the measure ranges from 0-48, with higher scores indicating greater severity of opioid withdrawal signs and symptoms.
Opioid-related Craving | 3 months post-randomization
  Mean change in self-reported opioid craving scores on the five-item Penn Craving Scale (PCS). Total scores on this measure range from 0 - 30, with higher scores indicating more severe craving for opioids.
Overall Quality of Life and General Health | 3 months post-randomization
  Mean change in self-reported Overall Quality of Life and General Health domain scores using the United States version of the World Health Organization (WHO) Quality of Life Scale - Brief. Participants rate items using a five-point Likert scale ranging from Not at all (1) to Completely (5). Raw scores within this domain range from 2-10. Higher scores indicate a higher overall quality of life and general health.
Physical Health | 3 months post-randomization
  Mean change in self-reported Physical Health domain scores using the United States version of the WHO Quality of Life Scale - Brief. Participants rate items using a five-point Likert scale ranging from Not at all (1) to Completely (5). Raw scores within this domain range from 7-35. Higher scores indicate a higher quality of physical health.
Psychological Health | 3 months post-randomization
  Mean change in self-reported Psychological domain scores using the United States version of the WHO Quality of Life Scale - Brief. Participants rate items using a five-point Likert scale ranging from Not at all (1) to Completely (5). Raw scores within this domain range from 6-30. Higher scores indicate a higher quality of psychological health.
Quality of Social Relationships | 3 months post-randomization
  Mean change in self-reported Social Relationships domain scores using the United States version of the WHO Quality of Life Scale - Brief. Participants rate items using a five-point Likert scale ranging from Not at all (1) to Completely (5). Raw scores within this domain range from 3-15. Higher scores indicate a higher quality of social relationships.
Quality of Environment | 3 months post-randomization
  Mean change in self-reported Environment domain scores using the United States version of the WHO Quality of Life Scale - Brief. Participants rate items using a five-point Likert scale ranging from Not at all (1) to Completely (5). Raw scores within this domain range from 8-40. Higher scores indicate a higher quality of environment.
Recovery Capital | 3 months post-randomization
  Mean change in self-reported recovery capital scores on the Brief Assessment of Recovery Capital - 10 (BARC-10). Scores on this measure range from 6-60, with higher scores indicating greater recovery capital and a higher likelihood of sustaining recovery from substance use disorder.
Depression Symptom Severity | 3 months post-randomization
  Mean change in self-reported depression symptom severity as measured by the Patient Health Questionnaire - 9 (PHQ-9). Scores on this measure range from 0-27, with higher scores indicating more severe depression-related distress.
Anxiety Symptom Severity | 3 months post-randomization
  Mean change in self-reported depression symptom severity as measured by General Anxiety Disorder - 7 (GAD-7). Scores on this measure range from 0-21, with higher scores indicating more severe anxiety-related distress.
Blinding to Condition | 3 months post-randomization
  The proportion of participants randomized to the comparison group who believe that they were in the active tAN condition.

OTHER OUTCOMES:
Weekly PTSD Symptom Severity | Weekly for 3 months post-randomization
  Weekly ratings of self-reported PTSD symptom severity on the PTSD Checklist for DSM-5 (PCL-5). PCL-5 scores range from 0 - 80 with a higher score indicating more severe trauma-related distress due to PTSD symptoms.
Weekly Opioid Withdrawal Symptom Severity Self Rated | Weekly for 3 months post-randomization
  Weekly ratings of opioid withdrawal symptom severity on the Short Opiate Withdrawal Scale - Gossop (SOWS-Gossop). Participants rate each item on a scale ranging from 0 (None) to 3 (Severe). The total scale score ranges between 0 - 30, with higher scores indicating more severe withdrawal symptoms.
Weekly Opioid Withdrawal Symptom Severity Observer Rated | Weekly for 3 months post-randomization
  Weekly ratings of opioid withdrawal symptom severity on the Clinical Opiate Withdrawal Scale (COWS). The total score on the measure ranges from 0-48, with higher scores indicating greater severity of opioid withdrawal signs and symptoms.
Weekly Opioid-related Craving | Weekly for 3 months post-randomization
  Weekly ratings of self-reported opioid-related craving on the PCS. Total scores on this measure range from 0 - 30, with higher scores indicating more severe craving for opioids.
Weekly Substance Use | Weekly for 3 months post-randomization
  Weekly non-prescribed substance use as indicated by Timeline Follow-back and urine drug test.
Bi-weekly Depression Symptom Severity | Bi-weekly for 3 months post-randomization
  Bi-weekly scores on the Patient Health Questionnaire - 9 (PHQ-9). Scores on this measure range from 0-27, with higher scores indicating more severe depression-related distress.
Bi-weekly Anxiety Symptom Severity | Bi-weekly for 3 months post-randomization
  Bi-weekly scores on the General Anxiety Disorder - 7 (GAD-7). Scores on this measure range from 0-21, with higher scores indicating more severe anxiety-related distress.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Sprunger, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- Gibson Center for Behavioral Change, Cape Girardeau, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We will create a completely de-identified dataset to prevent linkages to individual research participants. This includes removal of all Protected Health Information (PHI) and indirect identifiers that are not listed as PHI but could lead to "deductive disclosure" such as site numbers.
  Proprietary protocols regarding the Sparrow device are the intellectual property of Spark Biomedical, Inc. and will not be shared.
  This dataset, with related study materials (e.g., study protocol, define file, data dictionary, etc.), will be made available to investigators with a data-sharing agreement. The data sharing agreement will require commitment to: 1) not re-disclose the data; 2) secure the data; 3) use the data for research purposes only; 4) make no attempt to identify individual participants; 5) destroy the data once the planned research activities have been completed; and 6) follow all relevant National Institutes of Health (NIH) policies.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The shared data will be made available to other users by no later than the main findings are accepted for publication or 1-year post-study completion, whichever comes first. Published studies will have their own subcollections in the master Open Science Framework (OSF) project collection with the exact dataset used for the manuscript. These subcollections will have DOIs to aid in findability. We will include the DOI in relevant publications. The de-identified data will be retained indefinitely.
Access Criteria: Data will be findable for the research community through the OSF collection that will be established when this application is funded. We will reference the shared data in OSF in peer-reviewed publications and relevant webpages. For each publication, an OSF subcollection will be created within the master OSF project. Each subcollection will have a digital object identifier (DOI) associated with it. This data DOI will be referenced in the publication and associated presentations to allow the research community easy access to the exact data used in the publication. When these links are followed, researchers will view the instructions and requirements for establishing a data use agreement for access.
  Access to the data will be controlled and require a signed data use agreement. PI Sprunger will be responsible for administering these agreements.